CLINICAL TRIAL: NCT00489775
Title: Duloxetine Versus Paroxetine in the Acute Treatment of Major Depression
Brief Title: Duloxetine Versus Paroxetine for Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6937; F1J-AA-HMCV
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Duloxetine
Drug: Paroxetine

SUMMARY:
To determine if duloxetine works just as well as paroxetine in the treatment of major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* You are male or female at least 18 years of age with nonpsychotic major depression. Females of child-bearing potential must test negative on a pregnancy test at visit 1.

Exclusion Criteria:

* You have a serious medical illness, including any cardiovascular, hepatic, renal, respiratory, hematologic, endocrinologic, or neurologic disease, or clinically significant laboratory abnormality.
* You have a history of hepatic dysfunction, current jaundice, or positive hepatitis B surface Antigen or positive hepatitis C surface Antibody regardless of ALT.
* You have an ALT greater than or equal to 2 times the upper limit of normal.
* You have abnormal thyroid-stimulating hormone concentrations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2004-01; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To assess hypothesis that efficacy of duloxetine 60mg QD is non-inferior to paroxetine 20mg QD in treating major depressive disorder as defined by DSM-IV. Primary efficacy evaluated by mean change of HAMD17 total scores from baseline to endpoint.

SECONDARY OUTCOMES:
To compare the efficacy of duloxetine 60 mg QD and paroxetine 20 mg QD on anxiety symptoms associated with depression as measured by mean changes in Hamilton Anxiety Rating Scale (HAMA) total scores
To compare efficacy of treatment with duloxetine 60 mg QD and paroxetine 20 mg QD on symptoms of depression measured by mean endpoint scale on the Clinical Global Impression of Severity Scale (CGI-S) scale and the endpoint score
To compare efficacy of treatment with duloxetine 60 mg QD and paroxetine 20 mg QD on symptoms of depression measured by the endpoint score on the Patient Global Impression of Improvement (PGI-I) scale
To compare the efficacy of treatment with duloxetine 60 mg QD and paroxetine 20 mg QD on somatic complaints of pain as measured by the Somatic Symptom Inventory Scale (SSI) and Visual Analog Scales for pain (VAS)
To compare the efficacy of duloxetine 60 mg QD and paroxetine 20 mg QD as measured by response and remission rates
To compare the safety of duloxetine 60 mg QD and paroxetine 20 mg QD using information on treatment-emergent adverse events and other safety measures - e.g. electrocardiograms (ECGs) and laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing, China

REFERENCES:
- [Derived] Dodd S, Berk M, Kelin K, Zhang Q, Eriksson E, Deberdt W, Craig Nelson J. Application of the Gradient Boosted method in randomised clinical trials: Participant variables that contribute to depression treatment efficacy of duloxetine, SSRIs or placebo. J Affect Disord. 2014 Oct;168:284-93. doi: 10.1016/j.jad.2014.05.014. Epub 2014 Jun 4. PMID 25080392
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com